CLINICAL TRIAL: NCT00305929
Title: Phase II Study of Photodynamic Therapy With WST09 in Patients With Recurrent or Persistent Localized Carcinoma of the Prostate Following Radiation Therapy Failure - Repeat Procedure
Brief Title: Study of WST09 in Prostate Cancer After Radiation: Repeat Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: STEBA France (Industry)
Responsible Party: STEBA France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC/WST041251N/WST2.18
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Prostate Cancer
Keywords: Treatment of localized prostate cancer; Localized prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment with Tookad VTP
  Interventions: Drug: Treatment with Tookad VTP

INTERVENTIONS:
Drug: Treatment with Tookad VTP
  Other Names: WST09
Drug: Treatment with Tookad VTP — Tookad 2 mg/kg
Drug: Treatment with Tookad VTP — 2 mg/kg

SUMMARY:
This is a multi-centre, phase II, open-label, 12-month clinical trial for patients previously treated with WST09 (Tookad) who have positive prostate biopsies for cancer.

The study aims at delivering a second WST09 treatment for the purpose of eradicating the localized prostate cancer.

DETAILED DESCRIPTION:
Multi-centre, phase II, open-label, 12-month clinical trial for patients that previously received a vascular-targeted photodynamic treatment (VTP) with WST09 (Tookad) and still have histological findings (prostate biopsies) indicating the presence of localized cancer.

The WST09-mediated VTP procedure consists of an I.V. infusion of WST09 (Tookad) at 2 mg/kg, in combination with the per-cutaneous interstitial delivery of monochromatic laser light (of a wavelength of 763nm) via the trans-perineal implantation of illumination fibres, positioned in the prostatic lobes.

In a previous Tookad trial, escalating doses of laser light were used with a fixed dose of WST09 (2 mg/kg) in patients with localized prostatic cancer. Patients who underwent the procedure but still have positive prostate biopsies (residual cancer) may benefit from an additional WTS09-mediated VTP procedure. Thus, the aim of this study is to treat patients still presenting with localized prostate cancer with a second WST09-mediated VTP procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously treated with WST09-mediated VTP, with a positive biopsy of the prostate 6 months following treatment
* Disease confined to the prostate
* Life expectancy greater than 5 years

Exclusion Criteria:

* Unwilling or unable to give informed consent
* Patients who have received another treatment for their prostate cancer since their previous WST09-mediated VTP

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2006-03; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Prostate biopsy | 12 months

SECONDARY OUTCOMES:
MRI, PSA | 7 days, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Trachtenberg, MD, FRCS(C), Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- The Prostate Centre Princess Margaret Hospital, Toronto, Ontario, Canada